CLINICAL TRIAL: NCT02297373
Title: Clinical Predictors for Venous Thromboembolism in Patients With a History of Thrombosis
Brief Title: Clinical Predictors for Venous Thromboembolism in Patients With a History of Thrombosis (PREDICTORS)
Acronym: PREDICTORS
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20140622-01H
Record Dates: First submitted 2014-10-15; First posted 2014-11-21 (Estimated); Results first posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Thromboembolic Disease Recurrent; Deep Vein Thrombosis; Pulmonary Embolism; Venous Thromboembolism; Recurrent Thromboembolic Disease
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Venous Thromboembolism; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with a history of blood clots are at risk of developing additional clots in the future. Doctors use a tool called a clinical decision rule to tell them how likely it is that a patient has a blood clot and if they should have further testing to look for the clot. This tool may cause doctors to over-diagnosis a recurrent clot because the symptoms may be left over from the previous clot. Correctly diagnosing a recurrent blood clot is very important since there are risks associated with both over-diagnosis and under-diagnosis. If a recurrent blood clot is missed (under-diagnosis) the patient is at risk of death from a clot in the lungs. If blood thinners are prescribed when they are not needed (over-diagnosis), the patient may have to take blood thinners for their lifetime and risk having serious bleeding.

DETAILED DESCRIPTION:
Several tools have been developed to standardize the diagnostic management of a suspected first blood clot. One of these tools is the use of a clinical decision rule. Clinical decision rules have been designed to help clinicians make diagnostic and therapeutic decisions at the bedside. A score is computed on the presence of some criteria from the patient's medical history, clinical signs and symptoms. The score provides the probability of a blood clot. The rules can be used in combinations with a simple blood test - called D-dimer - to identify patients at low risk who don't require diagnostic imaging testing. Benefits include reduced costs, length in hospital and radiation exposure.

Patients with prior blood clots have been shown to be less likely to benefit from the non-invasive testing. Therefore, they often need to undergo imaging tests, which are frequently difficult to interpret in patients with prior blood clots since residual clots are often present and are difficult to distinguish from a recurrent clot.

The objective of this study is to try to prospectively assess the role of existing clinical decision rules in patients with prior blood clots, and to attempt to improve them in order to increase the yield of non-invasive testing and to reduce the risk of over-diagnosis with imaging tests.

With respect to this study, clots within the deep veins of the legs are called deep vein thrombosis (DVT), while clots in the lungs are called pulmonary embolism (PE).

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with clinically suspected acute recurrent DVT or PE regardless of whether the previous event was a DVT or PE
* Age ≥18 years old
* Willing and able to give informed consent

Exclusion Criteria:

* Life expectancy less than 3 months
* Suspicion of upper extremity thrombosis or thrombosis at an unusual site (e.g. cerebral or abdominal venous thrombosis)
* Previous VTE was distal DVT or subsegmental PE
* Suspected recurrent VTE is asymptomatic
* Previously enrolled in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients presenting with suspected acute recurrent venous thromboembolism (VTE).
Sampling Method: Non-Probability Sample
Enrollment: 744 (Actual)
Dates: Start 2014-11-19 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregoire Le Gal, MD, Principal Investigator — Ottawa Hospital
Locations (9):
- Canada (7):
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - Lawson Health Research Institute, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Hopital Montfort, Ottawa, Ontario
  - Humber River Hospital, Toronto, Ontario
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec
- Leiden University Medical Centre, Leiden, Netherlands
- Geneva University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mai V, Martens ESL, Righini M, Schulman S, Thiruganasambandamoorthy V, Kahn SR, Pecarskie A, Kovacs MJ, Visser S, Shivakumar S, Tan M, Kearon C, Rodger M, Scarvelis D, Delluc A, Girard P, Huisman MV, Wells PS, Klok FA, Le Gal G; PREDICTORS study group. Performance of clinical decision rules in patients presenting with suspected recurrent venous thromboembolism: a multicenter prospective cohort study. J Thromb Haemost. 2025 Oct;23(10):3239-3250. doi: 10.1016/j.jtha.2025.06.019. Epub 2025 Jun 25. PMID 40578691

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2014 to January 2019, eligible patients were recruited from six Canadian teaching hospitals, one academic center in Switzerland and one academic hospital in the Netherlands. All adult outpatients presenting to the Emergency Departments or Thrombosis Clinics of the participating hospitals with signs or symptoms suggestive of recurrent VTE and who were willing and able to give informed consent were eligible for inclusion.
Pre-assignment Details: Between Nov 2014 and Jan 2019, 744 participants consented and had baseline data and blood samples collected. Verification of prior VTE history excluded 21 with non-qualifying events, leaving 723 who met eligibility and were included. Those with recurrent VTE diagnosed at enrolment completed participation at the initial visit; those who did not have recurrent VTE diagnosed at enrolment were followed up by phone at Day 90.
Groups:
- Participant Eligibility: Of the 744 participants who provided informed consent and had baseline data and blood samples collected, 21 were later determined not to meet eligibility criteria after verification of prior VTE history (e.g., superficial vein thrombosis, below-knee DVT, subsegmental PE, or other non-qualifying events). These participants were excluded from analysis, leaving 723 who met all eligibility criteria and were included in the study.
Period: Overall Study
Arm/Group | Participant Eligibility
Started | 723
Completed | 705
Not Completed | 18

BASELINE CHARACTERISTICS:
Groups:
- Patients Presenting With Suspicion of Recurrent Venous Thromboembolism: Of the 744 participants consented, 723 met all eligibility criteria and were included in the study.
Arm/Group | Patients Presenting With Suspicion of Recurrent Venous Thromboembolism
Number analyzed (Participants) | 723
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 367
  Male | 356
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 657
  Black | 30
  Asian | 19
  Aboriginal | 10
  Hispanic | 2
  Caucasian and Aboriginal | 2
  Caucasian and Black | 2
  Caucasian and Asian | 1
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 29.6 (6.8)
Weight [Mean (Standard Deviation); unit: kilograms] | 87.6 (21.5)
Current Medication [Number; unit: participants]
  Aspirin | 104
  Clopidogrel | 11
  Anticoagulation | 322
  Oral estrogen therapy | 16
Type of Anticoagulation (n) [Count of Participants; unit: Participants] — Population: Of the 723 participants analyzed, 322 were currently taking an anticoagulant at the time of study inclusion
  Participants
    number analyzed (Participants) | 322
    Warfarin | 92
    Rivaroxaban | 124
    Dabigatran | 1
    Apixaban | 31
    Edoxaban | 1
    Low molecular weight heparin | 66
    Blinded study drug | 7
Known thrombophilia [Number; unit: participants] — Population: Of the 723 participants analyzed, 92 had known thrombophilia at the time of study inclusion. Participants could have more than one thrombophilia diagnosed.
  participants
    Antithrombin deficiency: number analyzed (Participants) | 92
    Antithrombin deficiency | 3
    Protein C deficiency: number analyzed (Participants) | 92
    Protein C deficiency | 8
    Protein S deficiency: number analyzed (Participants) | 92
    Protein S deficiency | 6
    Heterozygote Factor V Leiden: number analyzed (Participants) | 92
    Heterozygote Factor V Leiden | 46
    Homozygote Factor V Leiden: number analyzed (Participants) | 92
    Homozygote Factor V Leiden | 1
    Factor V Leiden unknown if heterozygote or homozygote: number analyzed (Participants) | 92
    Factor V Leiden unknown if heterozygote or homozygote | 5
    Prothrombin gene mutation: number analyzed (Participants) | 92
    Prothrombin gene mutation | 16
    Lupus anticoagulant: number analyzed (Participants) | 92
    Lupus anticoagulant | 8
    Anti-cardiolipins: number analyzed (Participants) | 92
    Anti-cardiolipins | 12
    Anti-Beta 2 glycoprotein 1: number analyzed (Participants) | 92
    Anti-Beta 2 glycoprotein 1 | 4
Family History of Venous Thromboembolism (VTE) [Count of Participants; unit: Participants]
  Yes | 213
  No | 510
Number of confirmed previous events [Count of Participants; unit: Participants] — Number of previous diagnostically confirmed events of venous thromboembolism prior to study inclusion
  Participants
    1 | 559
    2 | 130
    3 | 22
    4 | 10
    >/= 5 | 2
Type of last VTE event [Count of Participants; unit: Participants] — Breakdown of site of previously diagnosed venous thromboembolism (VTE). Of the 357 participants with a prior history of deep vein thrombosis (DVT, 12 were upper extremity DVT, 1 was concomitant upper and lower extremities DVT and 2 DVT of unknown location. Of the 79 participants that reported a prior history of pulmonary embolism (PE) and DVT, 1 participant had an upper extremity DVT. All other DVTs were in the lower extremity.
  Participants
    Pulmonary embolism (PE) | 237
    Deep vein thrombosis (DVT) | 357
    PE and DVT | 129
Active cancer [Number; unit: participants] | 79
Smoking status [Count of Participants; unit: Participants]
  Current smoker | 104
  Previous smoker | 227
  No smoking history | 392

OUTCOME MEASURES:

1. Primary Outcome: Validation of the Wells DVT Clinical Decision Rule
Description: The Wells DVT Clinical Decision Rule (CDR) assigns a score from -2 to +9 based on clinical variables (e.g., active cancer, limb swelling, localized tenderness, prior history of DVT, alternative diagnosis as likely or more likely than DVT). In this study, the 3-level Wells DVT CDR was applied prospectively at presentation (Day 0) to participants with suspected recurrent DVT, using data collected from patient history and physical examination. Scores classify patients into low (≤0), moderate (1-2), or high (≥3) probability of DVT. Higher scores indicate greater probability of recurrent DVT. The outcome measure was the rate of confirmed recurrent DVT events within each Wells category, confirmed by objective imaging and adjudicated by an independent committee.
Time Frame: Day 0 (at time of suspected recurrent DVT)
Population: Of the 723 participants included in the study, 401 presented with suspicion of isolated DVT, without signs or symptoms of PE. Of the 401 presenting with suspicion of isolated DVT, 108 had a confirmed diagnosis of DVT.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Presenting With Suspicion of Recurrent Venous Thromboembolism: A total of 744 participants provided informed consent. After verification of prior VTE history, 21 were excluded from analyses, leaving 723 in the study cohort. This outcome includes all participants assessed with the 3-level Wells DVT clinical decision rule at presentation for suspected recurrent DVT.
Arm/Group | Patients Presenting With Suspicion of Recurrent Venous Thromboembolism
Number analyzed (Participants) | 401
Participants
  Suspicion of Recurrent DVT: Score </= 0 (low) | 67
  Suspicion of Recurrent DVT: Score >/= 1-2 (moderate) | 186
  Suspicion of Recurrent DVT: Score >/= 3 (high) | 148
  Confirmed DVT during follow-up period: number analyzed (Participants) | 108
  Confirmed DVT during follow-up period: Score </= 0 (low) | 4
  Confirmed DVT during follow-up period: Score >/= 1-2 (moderate) | 39
  Confirmed DVT during follow-up period: Score >/= 3 (high) | 65

2. Primary Outcome: Validation of the Wells PE Clinical Decision Rule
Description: The 3-level Wells PE score (range 0-12.5) was calculated from history and exam at the index visit. Scores ≤4 = PE unlikely, >4 = PE likely. Higher scores indicate greater likelihood of PE. The outcome is the proportion with confirmed recurrent PE at the index diagnostic work-up, adjudicated by blinded review of imaging.
Time Frame: Day 0 (at time of suspected recurrent PE)
Population: Of the 723 participants enrolled, 268 presented with a suspicion of recurrent PE without concomitant DVT suspicion. Of the 268 presenting with suspicion of isolated PE, 79 had a confirmed diagnosis of PE.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Presenting With Suspicion of Recurrent Venous Thromboembolism: A total of 744 participants provided informed consent. After verification of prior VTE history, 21 were excluded from analyses, leaving 723 in the study cohort. This outcome includes all participants assessed with the 3-level Wells PE clinical decision rule at presentation for suspected recurrent PE.
Arm/Group | Patients Presenting With Suspicion of Recurrent Venous Thromboembolism
Number analyzed (Participants) | 268
Participants
  Suspicion of PE: Score <2 (low) | 83
  Suspicion of PE: Score 2-6 (moderate) | 160
  Suspicion of PE: Score >6 (high) | 25
  VTE recurrence confirmed during follow-up: number analyzed (Participants) | 79
  VTE recurrence confirmed during follow-up: Score <2 (low) | 11
  VTE recurrence confirmed during follow-up: Score 2-6 (moderate) | 56
  VTE recurrence confirmed during follow-up: Score >6 (high) | 12

3. Primary Outcome: Validation of the Geneva PE Clinical Decision Rule
Description: The revised Geneva score (range 0-22) was calculated from history and exam at the index visit. Scores 0-3 = low, 4-10 = intermediate, ≥11 = high probability. Higher scores indicate greater likelihood of PE. The outcome is the proportion with confirmed recurrent PE at the index diagnostic work-up, adjudicated by blinded review of imaging.
Time Frame: Day 0 (at time of suspected recurrent PE)
Population: Of the 723 participants included in the study, 268 presented with suspicion of PE, without signs or symptoms of DVT. Of the 268 presenting with suspicion of isolated PE, 79 had a confirmed diagnosis of PE.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Presenting With Suspicion of Recurrent Venous Thromboembolism: A total of 744 participants provided informed consent. After verification of prior VTE history, 21 were excluded from analyses, leaving 723 in the study cohort. This outcome includes all participants assessed with the revised Geneva PE clinical decision rule at presentation for suspected recurrent PE.
Arm/Group | Patients Presenting With Suspicion of Recurrent Venous Thromboembolism
Number analyzed (Participants) | 268
Participants
  Suspicion of recurrent PE: Score 0-3 (low) | 46
  Suspicion of recurrent PE: Score 4-10 (intermediate) | 181
  Suspicion of recurrent PE: Score >/= 11 (high) | 41
  Confirmed diagnosis of PU: number analyzed (Participants) | 79
  Confirmed diagnosis of PU: Score 0-3 (low) | 2
  Confirmed diagnosis of PU: Score 4-10 (intermediate) | 56
  Confirmed diagnosis of PU: Score >/= 11 (high) | 21

4. Secondary Outcome: Accuracy of Current D-dimer Testing Methods
Description: D-dimer testing at the index visit was performed using the institutional cut-off for positivity in place during the study period (2014-2019). Results were classified as positive or negative. The outcome is the proportion with confirmed recurrent VTE in each test category at the index diagnostic work-up, adjudicated by blinded review of imaging.
Time Frame: Day 0 (at time of suspected recurrent VTE)
Population: Of the 723 participants in the study cohort, the attending physician ordered D-dimer testing in 482 at presentation for suspected recurrent VTE. This outcome measure is based on the 169 participants from that group who had negative D-dimer results and were evaluated for recurrent VTE.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Presenting With Suspicion of Recurrent Venous Thromboembolism: A total of 744 participants provided informed consent. After verification of prior VTE history, 21 were excluded from analyses, leaving 723 in the study cohort. This outcome includes the 169 cohort participants with a negative D-dimer result at the index visit for suspected recurrent VTE.
Arm/Group | Patients Presenting With Suspicion of Recurrent Venous Thromboembolism
Number analyzed (Participants) | 169
Participants
  Negative D-dimer with recurrent VTE diagnosed | 6
  Negative D-dimer with no recurrent VTE diagnosed | 163

5. Secondary Outcome: Rate of Confirmed Events Using Current Wells DVT/Wells PE/Geneva PE in Participants on Anticoagulant Therapy
Description: The Wells DVT, Wells PE, and Geneva PE scores were calculated at the index visit in participants on anticoagulation. Score ranges and cut-offs as per respective rules. The outcome is the proportion with confirmed recurrent VTE in each risk category at the index diagnostic work-up, adjudicated by blinded review of imaging.
Time Frame: Day 0 (at time of suspected recurrent VTE)
Population: Of the 723 participants included, 38 were receiving anticoagulant therapy at the time of study inclusion and had a confirmed recurrent VTE. Of the 38 confirmed recurrent VTE events, 27 were for recurrent DVT and 11 were recurrent PE.
Measure: Count of Participants; unit: Participants
Groups:
- Patients Presenting With Suspicion of Recurrent Venous Thromboembolism: A total of 744 participants provided informed consent. After verification of prior VTE history, 21 were excluded from analyses, leaving 723 in the study cohort. This outcome includes participants who were receiving anticoagulant therapy at the index visit and underwent assessment with the Wells DVT, Wells PE, or revised Geneva PE clinical decision rules.
Arm/Group | Patients Presenting With Suspicion of Recurrent Venous Thromboembolism
Number analyzed (Participants) | 38
Participants
  Patients on anticoagulation with confirmed DVT using 3-level Wells Score: number analyzed (Participants) | 27
  Patients on anticoagulation with confirmed DVT using 3-level Wells Score: Low | 1
  Patients on anticoagulation with confirmed DVT using 3-level Wells Score: Moderate/Intermediate | 9
  Patients on anticoagulation with confirmed DVT using 3-level Wells Score: High | 17
  Patients on anticoagulation with confirmed PE using 3-level Wells Score: number analyzed (Participants) | 11
  Patients on anticoagulation with confirmed PE using 3-level Wells Score: Low | 1
  Patients on anticoagulation with confirmed PE using 3-level Wells Score: Moderate/Intermediate | 7
  Patients on anticoagulation with confirmed PE using 3-level Wells Score: High | 3
  Patients on anticoagulation with confirmed PE using revised Geneva Score: number analyzed (Participants) | 11
  Patients on anticoagulation with confirmed PE using revised Geneva Score: Low | 0
  Patients on anticoagulation with confirmed PE using revised Geneva Score: Moderate/Intermediate | 10
  Patients on anticoagulation with confirmed PE using revised Geneva Score: High | 1

6. Secondary Outcome: All-Cause Mortality Within 90 Days of Index Visit
Description: Number of participants who died from any cause from enrollment (Day 0) through Day 90 follow-up for those without confirmed recurrent VTE at enrollment.
Time Frame: From enrollment (Day 0) through Day 90 follow-up for those not diagnosed with a confirmed recurrent VTE at enrollment
Measure: Count of Participants; unit: Participants
Groups:
- All-cause Mortality for Patients Who Did Not Have Recurrent VTE Confirmed at Enrollment: A total of 744 participants provided informed consent. After verification of prior VTE history, 21 were excluded from analyses, leaving 723 in the study cohort. This outcome includes all-cause deaths recorded from Day 0 through Day 90 follow-up, unless diagnosed with a confirmed recurrent VTE at baseline.
Arm/Group | All-cause Mortality for Patients Who Did Not Have Recurrent VTE Confirmed at Enrollment
Number analyzed (Participants) | 723
Participants | 9

ADVERSE EVENTS:
Time Frame: From enrollment (Day 0) through Day 90 follow-up for participants not diagnosed with a confirmed recurrent VTE at enrollment.
Description: This was an observational diagnostic study with no investigational intervention. No adverse events were systematically collected. Per protocol, only all-cause mortality was assessed as a predefined secondary outcome. All deaths are reported in the All-Cause Mortality AE table below. The Serious and Other Adverse Event tables are completed with 0 events, as no additional adverse events were monitored.
Groups:
- All-cause Mortality: Participants that died of any cause from time of enrolment through the 90 day follow-up period.
Arm/Group | All-cause Mortality
All-Cause Mortality (participants affected / at risk) | 12/723
Serious Adverse Events (participants affected / at risk) | 0/723
Other Adverse Events (participants affected / at risk) | 0/723

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT02297373/Prot_SAP_000.pdf